CLINICAL TRIAL: NCT07108218
Title: Lateral Positioning During the Anesthesia Emergence After Ambulatory Adenotonsillectomy in Children on Postoperative Respiratory Adverse Events: a Multi-center Randomized Controlled Trial
Brief Title: Lateral Positioning for Extubation After Adenotonsillectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Peng Liang，MD, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025HX880
Record Dates: First submitted 2025-07-06; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Respiratory Adverse Events; Adenoidectomy; Tonsillectomy; Children
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Given the intervention's nature, full blinding was impossible; only postoperative data collectors and analysts were blinded. To minimize potential bias, we plan to maintain blinding among participants, anesthesiologists and surgeons in the operating room, the data collectors who conduct inpatient and telephone follow-up visits and data analysts. However, blinding could not be preserved for investigators, post-anesthesia care unit (PACU) outcome measure recorders, care providers in the PACU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral position group (Experimental): In the experimental group, the children will be placed in a head-up 30° lateral position for tracheal extubation and observation at the end of the procedure.
  Interventions: Procedure: lateral postion
- the supine position group (Placebo Comparator): In the control group, the patients will be placed into a supine position for extubation and observation at the end of the procedure.
  Interventions: Procedure: supine position

INTERVENTIONS:
Procedure: lateral postion — The children will be positioned on their sides with their heads elevated by 30°, a thin pillow behind their backs, the upper legs bent, and the lower legs straightened.
  Arms: lateral position group
Procedure: supine position — The children will be changed to a supine flat-lying position for extubation.
  Arms: the supine position group

SUMMARY:
The postoperative recovery period following general anesthesia has been associated with a 30%-50% incidence of postoperative respiratory adverse events (PRAEs) in pediatric populations, including laryngospasm, airway obstruction, and hypoxemia. Despite the limited effects of existing pharmacological and operative interventions, positional optimization (e.g., lateral or semirecumbent position) may play a potential role by decreasing airway resistance and improving oxygenation. However, evidence-based evidence for its use in pediatric populations is still lacking, necessitating the urgent need for randomized controlled trials.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, RCT conducted at four tertiary hospitals in China. It will be planned to include 350 subjects who meet the inclusion criteria and will be randomly divided into the lateral position and supine position group in a 1:1 ratio by the method of block group randomization stratified by centers. In the supine position group, the children will be extubated at the end of the procedure and observed in the decubitus position until the patient's Aldrete score was >9 and they left the PACU, whereas in the lateral position group, the children will be extubated and observed in the head-up 30° lateral position. The primary outcome is the incidence of PRAEs. Secondary outcomes included frequency of PRAE, number of airway devices used during the postoperative recovery period, time to tracheal extubation, length of stay in the recovery room, and incidence of PRAE at 24 hours and 7 days. postoperatively. Safety outcomes include the incidence of peripheral IV access dislodgement, monitoring device detachment rate, and patient falls rate. Exploratory outcomes comprise pain levels (assessed via the FLACC scale), agitation scores (PAED scale), sedation scores (Ramsay scale), and PONV scores, all evaluated at postoperative extubation and PACU discharge.

ELIGIBILITY:
Inclusion criteria:

1. Subjects aged 1-6 years old without gender limit.
2. Scheduled for an ambulatory adenotonsillectomy under general anesthesia.
3. American Society of Anesthesiologists (ASA) classification grade I or II.
4. Informed consent obtained from the patients' parents or legal guardians, who have expressed willingness to cooperate.

Exclusion criteria:

1. Presence of concomitant cardiac or pulmonary dysfunction or other significant systemic comorbidities.
2. History of difficult airway management or congenital/acquired structural anomalies of the airway.
3. Active respiratory tract infection within 30 days preceding surgery.
4. Preoperative neurological disorders or developmental abnormalities.
5. Intraoperative occurrence of major complications necessitating deviation from the planned anesthesia protocol or surgical procedure.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
the occurrence of postoperative respiratory adverse events (PRAEs) | during PACU
  PRAEs include a diverse array of respiratory complications, including laryngospasm, bronchospasm, apnea, airway obstruction, stridor, cough/choking, hypoxemia.

SECONDARY OUTCOMES:
Frequency of PRAEs | during PACU
  Frequency of PRAEs: Record the category and count of each PRAE occurring in each child.
Number of Emergency Airway Interventions | during PACU
  Number of Emergency Airway Interventions: including verbal stimulation, abdominal comparession, jaw thrust, mask ventilation, rescue intubation, etc
Tracheal extubation time | during PACU
  Tracheal extubation time: From the time the patient is transferred to the PACU until the intubation is removed. Extubation criteria: spontaneous breathing recovery and spontaneous eye opening.
PACU stay duration | during PACU
  PACU stay duration: time from PACU admission until meeting PACU discharge criteria(*Aldrete score ≥9/10)
Length of hospital stay | postoperative day 1
  Length of hospital stay
The PRAEs at 24 hours after surgery | at 24 hours postoperatively
  The PRAEs at 24 hours after surgery include laryngospasm, bronchospasm, airway obstruction, stridor, cough/choking, hypoxemia, upper respiratory tract infection and pulmonary infection.
The PRAEs at 7 days after surgery | at 7 days postoperatively
  The PRAEs at 7 days postoperatively include laryngospasm, bronchospasm, airway obstruction, stridor, cough/choking, hypoxemia, upper respiratory tract infection and pulmonary infection.

OTHER OUTCOMES:
Adverse events | during PACU
  Adverse events include the incidence of peripheral intravenous access dislodgment, monitoring device detachment rate, and the rate of bed falls. Other adverse events including hypertension, hypotension, tachycardia, bradycardia, arrhythmias are also recorded.
Pain score | every 10 minutes after extubation, when leaving the PACU.
  Pain levels are evaluated using the FLACC scale. The scale has 5 categories (face, legs, activity, cry, consolability). Each category is scored on the 0-2 scale, which results in a total score of 0-10 (0=relaxed and comfortable; 1-3=mild discomfort; 4-6 = moderate pain; 7-10 = sever discomfort or pain or both).
Emergence agitation | every 10 minutes after extubation, when leaving the PACU.
  Emergence agitation are evaluated using the PAED scale defined as a score ≥10.
Sedation scores | every 10 minutes after extubation, when leaving the PACU.
  Sedation scores are evaluated using the Ramsay scale. The Ramsay sedation score with scores of 1(irritability), 2(consciousness and cooperative), 3(deeper sleep and more agile response), 4(lighter sleep with faster awakening time), 5(sound sleep with slow response), and 6(no response) points, respectively.
Postoperative nausea and vomiting (PONV) | every 10 minutes after extubation, when leaving the PACU.
  The assessment of postoperative nausea and vomiting (PONV) involves observing and inquiring about the presence of nausea, vomiting, or retching in the child.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No